CLINICAL TRIAL: NCT00227162
Title: Pilot Study of Changing Exercise and Physical Activity Behavior in Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary E. Charlson, MD, Principal Investigator, Weill Medical College of Cornell University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N01-HC-25196 (0103-661); N01HC25196 (NIH)
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: Asthma; Behavior change; Physical activity; Risk reduction
MeSH Terms: conditions — Asthma; Motor Activity; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Active Comparator): Positive affect
  Interventions: Behavioral: Group 1
- Group 2 (Active Comparator): Self-Affirmation
  Interventions: Behavioral: Group 2
- Group 3 (Active Comparator): Positive Affect and self-affirmation
  Interventions: Behavioral: Group 3
- Group 4 (No Intervention): Control group

INTERVENTIONS:
Behavioral: Group 1 — Patients set a physical activity goal and were assigned to one of four groups. Patients were assigned to receive positive affect intervention.
  Other Names: Positive Affect; Control
  Arms: Group 1
Behavioral: Group 2 — Patients set a physical activity goal and were assigned to one of four groups. Patients were assigned to receive the self-affirmation intervention.
  Other Names: Self-affirmation
  Arms: Group 2
Behavioral: Group 3 — Patients set a physical activity goal and were assigned to one of four groups. Patients were assigned to receive both positive affect and self-affirmation intervention.
  Other Names: Positive Affect and Self-Affirmation
  Arms: Group 3

SUMMARY:
The objective of this pilot study is to assess the feasibility and the potential differential impact of a novel intervention of induced positive affect and self-affirmation to increase physical activity in asthma patients.

DETAILED DESCRIPTION:
The goals of this pilot study are to empirically test different interventional approaches to induce positive affect and self-affirmation. At the start of the study all patients in conjunction with their physicians will select a program of mild to moderate physical activity or exercise to be adopted and maintained on a routine basis. Patients also will complete the Paffenbarger Physical Activity and Exercise Index. Patients then will be divided into four groups according to the intervention they receive: 1) positive affect; 2) self-affirmation; 3) positive affect and self-affirmation; 4) control. The main outcome is the change in the Paffenbarger Physical Activity and Exercise Index scores from enrollment to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for this study if their physicians consider them medically able to participate, if they are 18 years of age or older, and if they have a diagnosis of mild to moderate asthma based on the NHLBI Asthma Expert Panel's classification system which rates symptoms, frequency of exacerbations, nocturnal attacks, activity restriction, use of medications, and pulmonary function.

Exclusion Criteria:

Patients will be excluded from this study for the following reasons:

* If they are unable to walk several blocks for whatever reason;
* If they have musculoskeletal or neurological deficits that preclude increased physical activity;
* If they have other pulmonary diseases;
* If they have cardiac disease or other severe comorbidity;
* If they are unable to provide informed consent because of cognitive deficits;
* If they refuse to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-02; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Change in Paffenbarger Physical Activity and Exercise Index scores from enrollment to 4 weeks. | 1-2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mancuso, MD, Principal Investigator — Weill Medical College of Cornell University; Mary E Charlson, MD, Study Director — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No Plan to Share IPD

REFERENCES:
- [Background] Mancuso CA, Rincon M, McCulloch CE, Charlson ME. Self-efficacy, depressive symptoms, and patients' expectations predict outcomes in asthma. Med Care. 2001 Dec;39(12):1326-38. doi: 10.1097/00005650-200112000-00008. PMID 11717574
- [Background] Mancuso CA, Peterson MG. Different methods to assess quality of life from multiple follow-ups in a longitudinal asthma study. J Clin Epidemiol. 2004 Jan;57(1):45-54. doi: 10.1016/S0895-4356(03)00248-8. PMID 15019010
- [Background] Mancuso CA, Peterson MG, Charlson ME. Comparing discriminative validity between a disease-specific and a general health scale in patients with moderate asthma. J Clin Epidemiol. 2001 Mar;54(3):263-74. doi: 10.1016/s0895-4356(00)00307-3. PMID 11223324
- [Background] Mancuso CA, Rincon M, Charlson ME. Adverse work outcomes and events attributed to asthma. Am J Ind Med. 2003 Sep;44(3):236-45. doi: 10.1002/ajim.10257. PMID 12929143
- [Background] Mancuso CA, Peterson MG, Charlson ME. Effects of depressive symptoms on health-related quality of life in asthma patients. J Gen Intern Med. 2000 May;15(5):301-10. doi: 10.1046/j.1525-1497.2000.07006.x. PMID 10840265